CLINICAL TRIAL: NCT02956954
Title: Follow-up of Myocardial T1 Relaxation Time in Patients With Anderson Fabry Disease (AFD): Impact of Treatment by Agalsidase Alpha (Replagal®)
Brief Title: Follow-up of Myocardial T1 Relaxation Time in Patients With Anderson Fabry Disease
Acronym: MyFABT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/092/HP
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anderson-Fabry Disease
Keywords: Enzyme replacement therapy
MeSH Terms: conditions — Fabry Disease | interventions — Enzyme Replacement Therapy; alpha-Galactosidase; agalsidase alfa; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient treated with Enzyme replacement therapy (Experimental): Magnetic Resonance Imaging will be done every 6 months for patient treated with Enzyme replacement therapy (Agalsidase alpha (Replagal®))
  Interventions: Drug: Enzyme replacement therapy (Agalsidase alpha (Replagal®)); Procedure: Magnetic Resonance Imaging
- Patient no treated with Enzyme replacement therapy (Sham Comparator): Magnetic Resonance Imaging will be done every 6 months for patient treated with Enzyme replacement therapy (Agalsidase alpha (Replagal®))
  Interventions: Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Enzyme replacement therapy (Agalsidase alpha (Replagal®)) — Patient treated with Enzyme replacement therapy as usual (Agalsidase alpha (Replagal®)). The treatment is prescribed in routine and not specially for the protocol
  Arms: Patient treated with Enzyme replacement therapy
Procedure: Magnetic Resonance Imaging — Magnetic Resonance Imaging will be assessed every 6 months during 2 years

SUMMARY:
Anderson Fabry disease (AFD) is an X-linked lysosomal storage disorder caused by a deficiency of the enzyme alpha-galactosidase. AFD can involve various organs and lead to a series of clinical abnormalities. Left ventricular hypertrophy in middle-aged men is one of its life threatening complications. It was shown that pending the absence of myocardial replacement fibrosis, substitution therapy could improve myocardial morphology and function as well as exercise capacity. Today, there is no available marker of the efficacy of the treatment on the heart morphology and function.

The T1 time (or longitudinal relaxation time) is one of the major components of the image formation in Magnetic Resonance Imaging (along with T2 time and proton density). Several techniques have been described to assess the myocardial T1-time.

One of them called MOLLI (Modified Look Locker Inversion Recovery), was made available in research centres by the Siemens company. In a study published in 2013, Sado et al. showed in a series of various conditions (hypertension, AFD, hypertrophic cardiomyopathy, AL amyloidosis, aortic stenosis and healthy volunteers) that a septal T1 below a threshold of 940ms could discriminate AFD patients. No overlap was shown with other conditions in this study. Our experience with T1 mapping supports that finding (even though our threshold could be slightly different), and we could recently detect by MRI a number of AFD patients, some of them with hypertrophy, some others without hypertrophy. The effect of Replagal® on the T1 relaxation time remains unknown.

The purpose of that study was to follow-up the heart morphology, function and myocardial T1 relaxation time in a population of treated/untreated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with proven Anderson Fabry Disease
* Patient with no Agalsidase alpha (Replagal®) treatment or
* Patient with Agalsidase alpha (Replagal®) treatment ongoing

Exclusion Criteria:

* Pace Maker / Implantable Cardiac Defibrillator
* Claustrophobia
* Ocular foreign body
* Allergy to gadolinium chelates
* Pregnancy ongoing
* Age < 18 years l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Difference from baseline in Septal myocardial T1 relaxation time | 24 months
  Septal myocardial T1 relaxation time will be evaluated using MRI for treated and untreated patient

SECONDARY OUTCOMES:
Difference from baseline in Septal myocardial T1 relaxation time | 6 months
  Septal myocardial T1 relaxation time will be evaluated using MRI for treated and untreated patient
Difference from baseline in Septal myocardial T1 relaxation time | 12 months
  Septal myocardial T1 relaxation time will be evaluated using MRI for treated and untreated patient
Difference from baseline in Septal myocardial T1 relaxation time | 18 months
  Septal myocardial T1 relaxation time will be evaluated using MRI for treated and untreated patient

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas DACHER, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No